CLINICAL TRIAL: NCT04666584
Title: Optimal Predilatation Treatment Before Implantation of a Magmaris Bioresorbable Scaffold In Coronary Artery Stenosis
Acronym: OPTIMIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Nørregaard Hansen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Odense University Hospital; S-20200114 (Other: Regional Committees on Health Research Ethics for Southern Denmark)
Record Dates: First submitted 2020-11-27; First posted 2020-12-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Stable Angina; Coronary Artery Stenosis; Myocardial Infarction; Cardiovascular Diseases; Myocardial Ischemia; Atherosclerosis of Artery; Coronary Disease; Heart Diseases; Arterial Occlusive Diseases
Keywords: bioresorbable scaffolds; optical coherence tomography; intravascular ultrasound; modified balloons
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Coronary Stenosis; Myocardial Infarction; Cardiovascular Diseases; Myocardial Ischemia; Coronary Disease; Heart Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Eligible patients randomized to predilatation with ScoreFlex balloon or a standard non-compliant balloon before percutaneous coronary intervention with implantation of a Magmaris bioresorbable scaffold.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Offline data analysis will be performed without knowing the allocated intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ScoreFlex balloon (Active Comparator): Pre-dilatation with a ScoreFlex balloon before implantation with a Magmaris bioresorbable scaffold
  Interventions: Device: ScoreFlex balloon
- Standard non-compliant balloon (Active Comparator): Pre-dilatation with a non-compliant balloon before implantation with a Magmaris bioresorbable scaffold
  Interventions: Device: Device: standard non-compliant balloon

INTERVENTIONS:
Device: ScoreFlex balloon — Pre-dilatation with a ScoreFlex balloon
  Arms: ScoreFlex balloon
Device: Device: standard non-compliant balloon — Pre-dilatation with a standard non-compliant balloon
  Arms: Standard non-compliant balloon

SUMMARY:
The aim of the study is to investigate if lesion preparation with a ScoreFlex balloon compared to a standard non-compliant balloon improve vascular healing and minimize lumen reduction after implantation of a Magmaris bioresorbable scaffold.

DETAILED DESCRIPTION:
Introduction: Ischemic heart disease (IHD) is characterized by progressive atherosclerosis in coronary arteries and may cause coronary artery stenosis or acute thrombus and occlusion. IHD is often treated with percutaneous coronary intervention (PCI) with balloon dilatation and implantation of a stent. The drug-eluting stents (DES) have been developed to minimize neointimal growth after implantation and reduce the risk of in-stent restenosis compared to bare-metal stents (BMS). Newer devices, bioresorbable scaffold (BRS), are made from a bioresorbable material slowly dissolving after implantation. The BRS guarantees optimal vessel support after balloon dilatation and implantation, but the artery can obtain original function and flexibility after the BRS has vanished. The development of the Magmaris BRS, with its improved radial strength, thinner struts compared to previous BRSs, is developed to reduce the complications seen in earlier generation BRS such as recoil, fracture and late stent thrombosis.

Previous studies have shown that coronary lesions treated with the previous generation of the Magmaris BRS resulted on lumen area reduction, possibly a consequence by increased plaque burden, compromising the scaffold area, combined with increased neointimal formation in the early phase of vascular healing and fast resolution.

Due to decreased radial strength of the BRS compared to metal stents, modification of plaque prior to BRS-implantation is necessary. The ScoreFlex balloon is a non-compliant balloon with circumference of fixated, scoring elements and permits controlled expansion and fragmentation of calcified plaque, compared to standard treatments with a non-compliant balloon.

Intravascular imaging with Intravascular Ultrasound (IVUS) and Optical Coherence Tomography (OCT) can assess the morphology and location of plaques in the coronary stenosis prior to PCI thereby optimizing the implantation. The scaffold-treated segment can also be evaluated with intravascular imaging components such as stent coverage, malapposition and neointimal hyperplasia, but only if the scaffold is visible. If the scaffold is dissolved, another method to assess the vascular healing is needed. IVUS can evaluate change in elastic external membrane (EEM), change in remodeling and minimal lumen area (MLA). The reduction in MLA is associated with increased neointimal hyperplasia and plaque burden in the vessel wall.

The aim of the study is to investigate if lesion preparation with a ScoreFlex balloon compared to a standard non-compliant balloon improve vascular healing and minimize lumen reduction after implantation of a Magmaris bioresorbable scaffold.

Method: The study is designed as a prospective randomized trial conduced at a single center (Odense University Hospital, Denmark). Eighty-two patients with stable angina pectoris and non-ST-segment elevation myocardial infarctions are included, if they meet the criteria. Pre-dilatation with a 2.0 mm balloon is performed followed by pre-interventional IVUS and OCT. Patients are randomized to lesion preparation and pre-dilatation with either the ScoreFlex balloon or a standard non-compliant balloon with a 1:1 balloon-to-artery ratio by measuring the reference segments. The residual stenosis should be less than 20 %. If the pre-dilatation goal is not achieved, up-scaling to a balloon 0,5 mm larger is allowed. The lesion is treated with implantation of a Magmaris scaffold. Finally, IVUS and OCT-images of the final result are obtained. Follow-up IVUS and OCT images are performed after 6 and 12 months.

Post-PCI OCT-images are analyzed at baseline and 6 and 12 months after index procedure. Change in MLA in the stented segment is measured with IVUS and OCT. The vascular healing is based on finding from the OCT images.

The study is submitted and approved by the Regional Committees on Health Research Ethics for Southern Denmark (Project-ID: S-20200114) and Danish Data Agency (Journal nr.: 20/49900) Statistics: Assuming data are normally distributed, categorical data will be presented as numbers and frequencies and compared using chi2-test. Continuous data will be presented as mean ± SD and compared using Student t-test- SPSS version 26.0 will be used for the statistical analysis.

The estimated sample size is based on data, from the HONEST study by Fallesen et al. The reduction of MLA from 6.99 mm2 to 5.01 mm (27%) 6 months after implantation of a Magmaris BRS, represented the expected reference group. Optimal lesion preparation with pre-dilatation with a ScoreFlex balloon is estimated to minimize MLA reduction from 6.99 mm2 to 6.22 mm2 (11%). A power calculation is conducted using the expected MLA after 6 months (6.22 mm2 for the ScoreFlex balloon and 5.01 mm2 for the standard non-compliant balloon). Inclusion of 35 patients in each group is necessary to reach statistical significance in case of 2-tailed significance level of 0.05 and power of 80 %. Loss to follow-up and poor image quality finalize an expected drop-out rate of 15 %, thereby requiring 82 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris and non-ST elevation myocardial infarction referred for invasive coronary angiography and percutaneous coronary intervention at Department of Cardiology, Odense University Hospital (Odense, Denmark)

Exclusion Criteria:

* participation in other randomized clinical trials
* life expectancy < 1 year
* allergy to aspirin, clopidogrel, ticagrelor or prasugrel
* eGFR < 30 mL/min
* tortuous and angiographically estimated extremely calcified lesions
* ostial, left main and bifurcation lesions
* lesions in a reference vessel diameter < 2.0 mm
* hemodynamic instability
* scheduled for coronary artery bypass grafting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-03-08 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Lumen Area | 6 months after index percutaneous coronary intervention
  Minimal Lumen Area

SECONDARY OUTCOMES:
Change in remodeling Index | 6 months and 12 months after index percutaneous coronary intervention
  Change in remodeling Index
Change in Minimal Lumen Area | 6 months and 12 months after index percutaneous coronary intervention
  Change in Minimal Lumen Area
Percentage of incomplete scaffold apposition | 6 months and 12 months after index percutaneous coronary intervention
  Percentage of incomplete scaffold apposition
Percentage of uncovered struts | 6 months and 12 months after index percutaneous coronary intervention
  Percentage of uncovered struts

CONTACTS AND LOCATIONS:
Overall Officials: Lisette O. Jensen, MD PhD Prof, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen KN, Maehara A, Troan J, Noori M, Hougaard M, Ellert-Gregersen J, Veien KT, Junker A, Hansen HS, Lassen JF, Jensen LO. Mechanistic insights into lumen reduction after implantation of a drug-eluting bioresorbable metallic scaffold assessed with serial intracoronary imaging: from the OPTIMIS trial. Coron Artery Dis. 2026 Mar 1;37(2):84-94. doi: 10.1097/MCA.0000000000001561. Epub 2025 Aug 20. PMID 40832681
- [Derived] Hansen KN, Troan J, Maehara A, Noori M, Hougaard M, Ellert-Gregersen J, Veien KT, Junker A, Hansen HS, Lassen JF, Jensen LO. Optimal Predilatation Treatment Before Implantation of a Magmaris Bioresorbable Scaffold in Coronary Artery Stenosis: The OPTIMIS Trial. Circ Cardiovasc Interv. 2025 Jan;18(1):e014665. doi: 10.1161/CIRCINTERVENTIONS.124.014665. Epub 2025 Jan 21. PMID 39836741